CLINICAL TRIAL: NCT05224778
Title: Assessing Pediatric Endpoints in DM1 (ASPIRE-DM1)
Brief Title: DMCRN-02-001: Assessing Pediatric Endpoints in DM1
Acronym: ASPIRE-DM1
Status: Recruiting | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM20023386
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Congenital Myotonic Dystrophy; CDM
Keywords: Clinical Research; Myotonic dystrophy; Congenital Myotonic Dystrophy; CDM
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and Tissue samples will be taken for biomarker development and retained for future research. No clinical diagnosis will be given to patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Congenital Myotonic Dystrophy (CDM): CDM group includes those aged neonate to 3 years, 11 months at enrollment. Individuals must have a diagnosis of CDM, which is defined as children having symptoms of myotonic dystrophy in the newborn period (<30 days), such as hypotonia, feeding or respiratory difficulty, requiring hospitalization to a ward or to the neonatal intensive care unit for more than 72 hours; and a genetic test confirming an expanded trinucleotide (CTG) repeat in the DMPK gene in the child or mother. An expanded CTG repeat size in the child is considered greater than 200 repeats or E1-E4 classification (E1= 200-500, E2=500-1,000, E3=1,000-1,500, E4>1,500).

SUMMARY:
The overall goal of the study is to establish valid clinical endpoint assessments for children with congenital myotonic dystrophy type 1 and develop biomarkers for the condition.

DETAILED DESCRIPTION:
Myotonic dystrophy type-1 (DM1) is an autosomal dominant disorder caused by a toxic CTG repeat expansion in the 3'UTR of the DMPK gene. DM1 is the most common adult-onset muscular dystrophy, with an overall prevalence of 1:8000. In approximately 10-20% of individuals with DM1, the onset of symptoms occurs at birth, which is known as congenital myotonic dystrophy (CDM).

Previous studies have enrolled a very limited number of children with CDM.

The rationale for this study is to include a larger population of patients with CDM in order to determine developmental milestones, measures of physical and cognitive function and quality of life, and correlate functional outcome measures with potential biomarkers in CDM .

ELIGIBILITY:
Inclusion Criteria:

* Age neonate to 3 years 11 months at enrollment.
* A diagnosis of CDM, which is defined as children having symptoms of myotonic dystrophy in the newborn period (<30 days), such as hypotonia, feeding or respiratory difficulty, requiring hospitalization to a ward or to the neonatal intensive care unit for more than 72 hours; and a genetic test confirming an expanded trinucleotide (CTG) repeat in the DMPK gene in the child or mother. An expanded CTG repeat size in the child is considered greater than 200 repeats or E1-E4 classification (E1= 200-500, E2=500-1,000, E3=1,000-1,500, E4>1,500).
* Guardian is willing and able to sign consent and follow study procedures

Exclusion Criteria:

* Any other non-DM1 illness that would interfere with the ability or results of the study in the opinion of the site investigator
* Significant trauma within one month
* Internal metal or devices (exclusion for DEXA component)
* History of bleeding disorder or platelet count <50,000
* History of reaction to local anesthetic

Max Age: 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 30 children with CDM
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-08-24 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate motor milestone attainment in individuals with CDM and ChDM and compare to typically developing children | Through study completion at 18 months
  Milestone Assessment using Peabody definitions: This survey would ask parents to assess the age of motor milestones in days, months of infant age. Birth history, including prematurity, ventilatory status, and feeding problems would also be collected on the CRF. Feeding and ventilatory support, as well as height and weight will be collected at each study visit.

SECONDARY OUTCOMES:
Dysarthria Assessment | Through study completion at 18 months
  A blinded, standardized video assessment tabulating language milestones by a trained rater will be conducted at each visit.
Vineland | Through study completion at 18 months
  The Vineland will be administered by an interviewer to ensure standardized intake of data. This assessment will capture the adaptive function, including gross motor and fine motor, as reported by the parent proxy.
CCMDHI | Through study completion at 18 months
  The congenital and childhood myotonic dystrophy health index is a disease specific patient or proxy reported outcome measure specific to these conditions. The current study will utilize the proxy version.
Domain Delta | Through study completion at 18 months
  This assessment asks parents for global impression of change related to the baseline visit and will be used as an anchoring measure for the statistical analyses.
Gross Motor Function Measure (GMFM-88) | Through study completion 18 months
  The GMFM assesses functional abilities like lying/rolling, sitting, crawling/kneeling, standing, and walking, running, and jumping.

OTHER OUTCOMES:
Correlate the functional outcome measures with potential biomarkers in CDM. | Baseline
  Fine needle muscle biopsy:On the baseline visit, a fine needle aspirate will be performed. Biopsy will only be peformed once to minimize the risk. The procedure will be performed with local anesthesia (1% lidocaine without epinephrine and free of preservatives) of the vastus lateralis. Following lidocaine injection, a fine needle will be used to aspirate the quadriceps muscle to obtain a total of one aspirate. The aspirate will be flash frozen in liquid nitrogen. A similar procedure has been performed on adults with DM1, and the average biopsy yields sufficient tissue for RNA-Seq analysis.
Blood Sampling | Baseline, month 12, month 18
  DNA and RNA samples will be processed by Virginia Commonwealth University.
Muscle mass, DEXA | Baseline, month 12, month 18
  Lean muscle mass will be evaluated using serial DEXA scans as an exploratory endpoint. All sites will use a Hologic DEXA scanner. Investigators will evaluate whole body lean mass, left and right arm lean mass, and left and right leg lean mass. Particularly early in childhood, investigators would expect rapid changes in lean muscle mass. If there were a divergence between controls and subjects with CDM, this would provide evidence that CDM is a disorder of muscle maturity, as well as provide a potential biomarker.
World Health Organization (WHO) Motor Milestones | Through study completion at 18 months
  The WHO Motor Milestones is a set of 6 standardized motor milestones that include 1) Sitting without support, 2) Standing with assistance, 3) Hands-&-knees crawling, 4) Walking with assistance, 5) Standing alone, and 6) Walking alone.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas E. Johnson, MD, Principal Investigator — Virginia Commonwealth University
Locations (5):
- United States (4):
  - University of California, Los Angeles, Los Angeles, California
  - University of Kansas Medical Center, Fairway, Kansas
  - University of Rochester Medical Center, Rochester, New York
  - Virginia Commonwealth University, Richmond, Virginia
- Centro Clinico NeMO, Milan, Italy

IPD SHARING:
Plan to Share IPD: No